CLINICAL TRIAL: NCT04416958
Title: Pacing for Cardiac Resynchronisation Using the Intrinsic Conduction System to Maintain Physiologic Ventricular Activation
Brief Title: Pacing to Maintain Physiologic Ventricular Activation
Acronym: Pace-Conduct
Status: Recruiting | Type: Observational
Sponsor: Klinikum-Fuerth (Other)
Collaborators: University of Erlangen-Nürnberg (Other); University of Trieste (Other)
Responsible Party: Sponsor
Other Study IDs: Pace_Cond_KHF
Record Dates: First submitted 2020-06-01; First posted 2020-06-04 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Pacemaker DDD; His Bundle Pacing; LBB Area Pacing; Pacing-Induced Cardiomyopathy; Left Bundle-Branch Block; ICD
Keywords: His bundle pacing; LBB area pacing; cardiac resynchronisation therapy
MeSH Terms: conditions — Bundle-Branch Block

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CIED for cardiac resynchronisation: Patients implanted with an CIED for cardiac resynchronisation aiming to avoid pacing induced ventricular dyssynchrony, e.g. His bundle pacing, LBB-area pacing, CRT. These different implanted types of devices may be further analysed as subgroups.
  Interventions: Device: cardiac implantable electronic device (CIED) implantation

INTERVENTIONS:
Device: cardiac implantable electronic device (CIED) implantation — CIED Implantation according to the Guidelines aiming to avoid pacing induced dyssynchrony

SUMMARY:
Right ventricular pacing causes ventricular dyssynchrony and may be associated with impaired outcome. In the last decade, several approaches for more physiological pacing became available and were implemented in the latest guidelines. However, compared to conventional device implantation, cardiac resynchronization, His bundle pacing and left bundle area pacing remain demanding procedures in the individual case. Goal of the single center observational "Pace conduct" study is to evaluate implantation success, safety and outcome of pacing methods that maintain physiologic ventricular activation.

DETAILED DESCRIPTION:
Background:

Conventional ectopic myocardial right ventricular pacing (RVP) causes ventricular dyssynchrony and may be associated with reverse ventricular remodeling, reduced ejection fraction (EF), left ventricular dilatation, functional mitral valve regurgitation, heart failure and an increased rate of new onset atrial fibrillation.

Dependent on individual patient's characteristics, several strategies are established to prevent and to overcome the potential drawbacks of chronic RVP. In general, unnecessary ectopic RVP should be avoided. For example, in patients with sinus node disease and intact atrioventricular (AV) conduction, atrial pacing, AV (search) hysteresis or AAI-DDD/ADI pacing may be used. In patients with impaired cardiac function and an expected higher percentage of RVP, pacing strategies for cardiac resynchronization are indicated. Conventional cardiac resynchronization therapy (CRT) uses an additional transvenous left ventricular lead for synchronous ventricular stimulation and was shown to shorten QRS duration and to reduce morbidity and mortality in patients with chronic heart failure, left bundle branch block (LBBB) and reduced EF. Due to the non-physiological left ventricular epicardial stimulation, however, conventional CRT is associated with 30% of non-responders and may even prolong ventricular activation in patients with narrower QRS complex. First described in 1968, His bundle pacing (HBP) has evolved to an increasingly used alternative for cardiac pacing. Currently, HBP is regarded the most physiologic approach for ventricular stimulation because it prevents ventricular dyssynchrony and its potential fatal long-term consequences by preserving normal electrical activation of the ventricles. Clinical benefit of HBP has been shown compared with conventional permanent RVP and CRT. Recent studies documented restoration of normal electrical and mechanical left ventricular synchrony for both selective and non-selective HBP. However, compared with conventional RVP the implantation procedure for HBP is much more demanding requiring exact placement of the pacing lead within the anatomically variable His bundle area. Alternatively, the correction of bundle branch conduction disorders has been demonstrated for left bundle branch area (LBBA) pacing. As a consequence, current guidelines recommend pacing methods that maintain physiologic ventricular activation in patients with atrioventricular block who have an indication for permanent pacing with a LVEF between 36% and 50% and are expected to require ventricular pacing more than 40% of the time (class IIa indication).

In summary, there is increasing evidence showing the benefits of the different strategies for physiologic pacing but the appropriate use of these approaches may be challenging in the individual case. Therefore, appropriate patient selection, implantation approaches, device programming and follow-up require further intensive evaluation.

Objective:

Main goal of the study is to evaluate implantation success for pacing methods aiming to maintain physiologic ventricular activation. Procedural success is defined as stable lead positioning and effective pacing within the target area with an appropriate and stable pacing threshold.

Secondary goals of the study are to document and to evaluate

* procedural parameters (e.g. venous access, time needed for lead implant, procedural duration, radiation) and adverse events dependent on procedural approaches and patients characteristics,
* performance of the implanted system (sensing, pacing thresholds) and clinical outcome during routine follow-up

Study design:

Single center, non-randomized, observational study, retrospective data analysis, on-going prospective patient enrollment, descriptive statistics.

Center: Klinikum Fuerth (Dept. for Heart and Lung diseases, section for clinical electrophysiology) / Germany in cooperation with the Dept. of Cardiology of the University Erlangen / Germany and the University of Trieste / Italy.

Patients and methods:

Primary endpoint: Implantation success. Effective pacing and acceptable pacing threshold at the targeted lead position. Target for lead placement is the area with maximum delayed ventricular activation for transvenous CRT, the His bundle for selective or non-selective HBP and the right interventricular septum with left bundle branch capture for LBBA pacing, respectively. Target thresholds for the lead placed within the coronary sinus or at the intrinsic conduction system is <2.5 V @ 1 ms with a maximum acceptable threshold of <4.0 V @ 2 ms or <5 V @ 1 ms. Target for all other leads is <1 V @ 0.5 ms.

Secondary endpoints: patient characteristics and association with outcome. Implantation success and outcome correlated with patient characteristics including electrocardiogram and echocardiographic parameter and procedure related techniques and parameter. Safety: radiation exposure, number and type of adverse events and adverse device related events. Follow-up: device function, interrogation, programming and clinical outcome as evaluated in routine follow-up, incl. ECG, echocardiography and parameter for assessment of heart failure. Subpopulations: managed ventricular pacing, His bundle pacing, LBB-area pacing, CRT. Implantation with or without electroanatomic mapping system.

Inclusion criteria:

Implantation of a pacemaker or ICD according to the current guidelines (Class I or IIa indication) aiming to avoid pacing induced dyssynchrony, e.g. managed ventricular pacing, His-bundle pacing, LBB-area pacing or conventional transvenous CRT. Age ≥ 18 years.

Exclusion criteria:

No given informed consent for the procedure. No follow up data available.

Sample size:

For the observational study, there is no pre-specified sample-size. Data from 200 patients and procedures are expected.

Data security:

Study related data are collected by the study investigators in an anonymous clinic-internal data-base that is password protected. All investigators have to provide valid GCP training.

Risk estimation:

The study is observational and descriptive with anonymized data collection and data analysis. Therefore, the study adds no risk to the study population.

Ethics:

The "Pace-Conduct" study has been approved by the responsible ethics committee of the Friedrich- Alexander University Erlangen, Germany (145_20 Bc)

ELIGIBILITY:
Inclusion Criteria:

* Pacemaker or ICD Implantation aiming to avoid pacing induced ventricular dyssynchrony according to current guidelines
* age >= 18 years

Exclusion Criteria:

* no informed consent for the procedure given
* no follow-up data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing Pacemaker or ICD Implantation according to current Guidelines with the aim to avoid pacing induced ventricular dyssynchrony.
  Subgroups according to type of device implanted, lead Position and programming.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
CIED Implantation success | peri-procedural
  successful Pacemaker- or ICD implantation with effective pacing and acceptable pacing threshold in the targeted area

SECONDARY OUTCOMES:
pre-operative: Implantation related Patient characteristics | 1 month post implantation
  association with procedural and post-implant outcome
intra-procedural: implant success related with procedural characteristics | peri-procedural
  correlation of Implantation success with Patient characteristics and procedural technical Parameter, eg. use of an electroanatomic mapping system
peri-procedural: safety and radiation | peri-procedural
  Radiation exposure and number and type of all adverse Events and adverse device associated events
follow-up: device function | one year
  device parameter and programming during follow up
follow-up: outcome | one year
  clinical Outcome during follow up

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Bastian, MD, Principal Investigator — Klinikum-Fuerth
Locations (1):
- Klinikum Fuerth, Fürth, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bastian D, Gregorio C, Buia V, Walaschek J, Rittger H, Vitali-Serdoz L. His bundle pacing guided by automated intrinsic morphology matching is feasible in patients with narrow QRS complexes. Sci Rep. 2022 Mar 4;12(1):3606. doi: 10.1038/s41598-022-07516-6. PMID 35246595